CLINICAL TRIAL: NCT02792647
Title: A Double-blind, Randomised, Placebo-controlled, Parallel Group, Dose Escalation Study to Investigate the Safety, Toleration, and Pharmacokinetics of Multiple Oral Doses of IX-01 in Healthy Male Subjects
Brief Title: A Study of Multiple Oral Doses of IX-01 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ixchelsis Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IX-0104
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Experimental: IX-01 (Experimental): 2 different dose groups 1,600 mg and 2,400 mg of IX-01 oral aqueous dispersion, administered once daily for 10 days
  Interventions: Drug: IX-01

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: IX-01 — Administered orally
  Arms: Experimental: IX-01

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of IX-01 after multiple doses, and to determine the PK of IX-01 and activity of CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

1. Male healthy volunteer.
2. Aged 18-45 years at the time of signing the informed consent.
3. A body mass index (Quetelet index) in the range 18-30.
4. Total body weight >50 kg at screening.
5. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
6. Willingness to comply with the contraception requirements of the trial.
7. Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
8. Willingness to give written consent to have data entered into The Overvolunteering Prevention System (TOPS).

Exclusion Criteria:

1. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer, including any of the following findings:

   * have lipid and/or liver function test results >1.25 x ULN or other clinical laboratory blood biochemistry test results outside the normal reference range unless discussed and approved by sponsor
   * history of unexplained syncope
   * family history of unexplained sudden death, or sudden death due to long QT syndrome
   * QTcF interval >450 msec in 2 of 3 consecutive ECGs (additional ECGs may be recorded, if required, but a median QTcF ≤ 450 msec from 3 consecutive ECGs is required for the volunteer to be considered eligible)
   * bundle branch block and other conduction abnormalities, other than mild first degree atrio-ventricular block
   * irregular rhythms other than sinus arrhythmia or occasional supraventricular ectopic beats
   * T-wave configuration of insufficient quality for determination of QT interval, as assessed by the investigator
2. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
3. Impaired gastrointestinal, endocrine, thyroid, hepatic, cardiovascular, respiratory, haematological, renal or neurological function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
4. Surgery (e.g. stomach bypass) or medical condition that might affect absorption of medicines.
5. Presence or history of severe adverse reaction to any drug.
6. Use of any prescription or over-the-counter medicine during the 14 days before the first dose of trial medication, or intention to use any medicine during the trial, with the exception of short courses of medication considered by the investigator not to interfere with the safety of the subject or the integrity of the trial data (such as acetaminophen (paracetamol)).
7. Current use of any herbal remedy or nutritional supplement, or intention to use any such product during the study.
8. Participation in another clinical trial of a new chemical entity or a prescription medicine within the 3 months prior to the first dose.
9. Previous participation in this trial or any other clinical trial of an oxytocin receptor antagonist.
10. Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly or more than 5 cigarettes daily.
11. Blood pressure and heart rate in supine position at the screening examination outside the ranges 90-130 mm Hg systolic, 50-90 mm Hg diastolic; heart rate 50-90 beats/min, unless judged not clinically significant by an investigator.
12. Possibility that the volunteer will not cooperate with the requirements of the protocol.
13. Evidence of drug abuse on urine testing.
14. Positive test for hepatitis B, hepatitis C or HIV1 or HIV2.
15. Loss of more than 400 mL blood during the 3 months prior to the first dose, eg as a blood donor.
16. Objection by General Practitioner (GP) to volunteer entering trial.
17. Employee of the investigator site or any company involved in sponsoring, organising or conducting the trial, or immediate family of the employee. Immediate family is defined as spouse, parent, child or sibling, whether biologically related or legally adopted.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Drug Related Adverse Events (AEs) or any Serious AEs | Baseline to Day 20 (Estimated up to 3 weeks)

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of IX-01 | Pre-dose to 24 hours post dose on Days 1 and 10
Area Under the Plasma Concentration-Time Curve (AUCtau) | Pre-dose up to 24 hours post dose on Days 1 and 10
Time of Peak Plasma Concentration (Tmax) of IX-01 | Pre-dose to 24 hours post dose on Days 1 and 10
Urine 6-β-hydroxycortisol/cortisol Ratio | Pre-dose on Day 1 and Day 10
Elimination Half Life (t1/2) of IX-01 | Pre-dose up to 96 hours post dose on Day 10
Accumulation Ratio (Racc) of IX-01 based on AUCtau | Pre-dose up to 24 hours post dose on Day 10
Accumulation Ratio (Racc) of IX-01 based on Cmax | Pre-dose up to 24 hours post dose on Days 1 and 10
Area Under the Concentration-Time Curve (AUCt) from Zero to the Time of Last Quantifiable Concentration (AUC(0-t)) of IX-01 | Pre-dose to 96 hours post dose on Day 10
Minimum Observed Concentration (Ctrough) of IX-01 | Pre-dose on Days 2 to 10
Elimination Rate Constant (Kel) of IX-01 | Pre-dose up to 96 hours post dose on Day 10
Apparent Clearance of IX-01 | Pre-dose up to 24 hours post dose on Day 10
Apparent Volume of Distribution During the Terminal Phase of IX-01 | Pre-dose up to 96 hours post dose on Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Franz van den Berg, MBChB, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No